CLINICAL TRIAL: NCT05563805
Title: Exploring Virtual Reality Adventure Training Exergaming (V-RATE) on Veterans' Health Outcomes
Brief Title: Exploring Virtual Reality Adventure Training Exergaming
Acronym: V-RATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Donna L. Schuman, Assistant Professor, The University of Texas at Arlington
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTexasArlington
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Physical Activity; Sedentary Behavior; Depression; Cognitive Function; Post Traumatic Stress Disorder; Quality of Life; Anxiety
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Depression; Stress Disorders, Post-Traumatic; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two group (intervention and control) randomized trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (Experimental): intervention participants will engage in a 30-minutes VR adventure games on a non-mobilized treadmill (5-min warm-up, 20-minutes treadmill, and 5-min cool-down) for a total of 6 sessions over 6-8 weeks. Participants in the V-RATE group will be instructed to self-pace walking/running on the treadmill while they are fully immersed in the VR games for two 10-minute bouts with a complete rest interval (heart rate reduces to normal range). Participants will complete measures at baseline, post-training, and one-month follow-up.
  Interventions: Device: Virtual Reality-based physical activity intervention
- Control (No Intervention): Control participants will not receive the intervention. Participants will complete measures at baseline, post-training, and one-month follow-up.

INTERVENTIONS:
Device: Virtual Reality-based physical activity intervention — The V-RATE intervention will be delivered through a 360-degree non-mobilized treadmill in a university clinical laboratory for 6-8-weeks (1-2 days/week, 30 minutes/session) totaling 6 sessions. The V-RATE program will be focused on creating a safe and immersive environment supportive of physical activity. The treadmill enables an individual can walk and run at self-paced speed, moving in 360-degrees (i.e., forwards, sideways, and backwards) without risk of falling. The core feature of the self-paced treadmill is a concave walking platform with an adjustable waist hardness that enables a safe, smooth, natural gait while adults with elevated BMI engage in an immersive walking and running motion. During the V-RATE intervention, participants will self-pace their locomotor action (walking/running/bending/ jumping) while they wear the VR headset and experience immersive VR adventure games using the Omniverse VR system.
  Arms: Intervention

SUMMARY:
The current project aims to design and implement an 8-week Virtual Reality Adventure Therapy Exergaming (V-RATE) intervention focused on women veterans. A randomized controlled trial using a repeated measure design with a 1-month follow-up assessment will be employed to examine effects on physical and mental health outcomes.

DETAILED DESCRIPTION:
The current project aims to design and implement an 8-week Virtual Reality Adventure Therapy Exergaming (V-RATE) intervention focused on veterans. A randomized controlled trial using a repeated measure design with a 1-month follow-up assessment will be employed. The project addresses two specific aims:

Aim 1. To examine the effects of an 8-week V-RATE intervention on physical health (i.e., BMI, physical activity, sedentary behavior) among veterans. We hypothesize that after controlling for socio-demographic variables and physical activity history, individuals in the V-RATE group would exhibit more improvement in the physical health indicators after the intervention compared to individuals in the control group. We further hypothesize gains would be maintained or enhanced at 1-month follow-up measure.

Aim 2. To examine the effects of an 8-week V-RATE intervention on mental health outcomes (i.e., depression, anxiety, posttraumatic stress, cognitive function, health-related quality of life), among veterans. We hypothesize that after controlling for socio-demographic variables and physical activity history, individuals in the V-RATE group will exhibit more improvement in the mental health indicators after the intervention compared to individuals in the control group. We further hypothesize gains maintained or enhanced at 1-month follow-up measure.

ELIGIBILITY:
Inclusion Criteria:

1. Are between the ages of 18 and 45
2. Identify as a U.S. military veteran

4. Normal vision (no colorblindness)

Exclusion Criteria:

1. Unable to walk independently (e.g., use of any mobility assistive device such as brace, wheelchair, cane, crutch, walker, knee scooter)
2. Self-reported joint problem that limits mobility (e.g., arthritis or other condition that would prevent participation) or ongoing orthopedic injury
3. Self-reported pregnancy or suspicion of pregnancy
4. Self-reported motor disorder or impaired sense of motion or balance (such as Parkinsonism)
5. Self-reported color blindness
6. Self-reported neurological or cognitive disorder (e.g., TBI, history of seizure)
7. Self-reported cardiac surgery or any ongoing cardiovascular issues preventing participation or physical activity.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female sex at birth
Enrollment: 40 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in depression from baseline to week 6-8 and one-month follow-up (Week 12) | Baseline, Week 6-8, Week 12
  Depression will be measured by self-report using the nine-item Patient Health Questionnaire-9 (PHQ-9).

SECONDARY OUTCOMES:
Anxiety change from baseline to week 6-8 and one-month follow-up (Week 12) | Baseline, post-training, Week 12
  Anxiety will be measured using the Beck Anxiety Inventory (BAI).
Posttraumatic Stress change from baseline to week 8 and one-month follow-up (Week 12) | Baseline, post-training, Week 12
  Posttraumatic Stress will be measured using the Posttraumatic Stress Disorder Checklist-5 (PCL-5).
Cognitive Function change from baseline to week 8 and one-month follow-up (Week 12) | Baseline, post-training, Week 12
  Cognitive Function will be measured via the Cambridge Neuropsychological Test Automated Battery (CANTAB) to assess the participants' executive function and working memory via multitasking test and spatial working memory tests.
Health-Related Quality of Life (HRQOL) change from baseline to week 8 and one-month follow-up (Week 12) | Baseline, Week 6-8, Week 24
  Health-Related Quality of Life (HRQOL) will be measured using the Short Form-36 Health Survey.
BMI change from baseline to week 6-8 and one-month follow-up (Week 12) | Baseline, post-training, Week 12
  Participants' height and weight will be measured to calculate their BMI.
Physical Activity and Sedentary Behavior change from baseline to week 8 and one-month follow-up (Week 12) | Baseline, Week 8, Week 24
  Physical Activity and Sedentary Behavior will be measured objectively using the ActiGraph GT9X accelerometers
Heart Rate Variability (SDNN, rMSSD, LF, HF) change from baseline to week 8 and one-month follow-up (Week 12) | Baseline, post-training, Week 12
  Heart Rate Variability will be measured using ECG (electrocardiogram)-derived heart rate variability from a Polar H10 Heart Rate Monitor Chest strap and HRV-monitoring app.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Arlington, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No